CLINICAL TRIAL: NCT04536207
Title: Effect of Cryotherapy in Controlling Peripheral Neuropathy in Cancer Children
Brief Title: Cryotherapy for Neuropathy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Lecturer of physical therapy, Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, South Valley University, Qena, Egypt., South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002570
Record Dates: First submitted 2020-08-16; First posted 2020-09-02 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Cancer
Keywords: Cancer; Peripheral neuropathy; Cryotherapy
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: They were assigned randomly into two equal groups.Group (A) study group received the same medical care and cryotherapy, three times / weak for three successful months. And group (B) control group received medical care and standard chemotherapy only.
Who Masked: Participant, Investigator
Masking Description: Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental): Group (A) the study group received cryotherapy
  Interventions: Other: Cryotherapy (apparatus)
- the control group (No Intervention): Group (B) the control group not received cryotherapy

INTERVENTIONS:
Other: Cryotherapy (apparatus) — Cryotherapy is a pain treatment that uses a method of localized freezing temperatures to deaden an irritated nerve. Cryotherapy is also used as a method of treating localized areas of some cancers (called cryosurgery), such as prostate cancer and to treat abnormal skin cells by dermatologists
  Arms: the study group

SUMMARY:
This study aimed to assess the efficacy of cryotherapy in controlling Peripheral Neuropathy in cancer children

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious condition characterized by symmetrical, distal damage to the peripheral nerves that may be caused by several classes of drugs, including chemotherapeutic agents. Chemotherapy-induced peripheral neuropathy (CIPN) is an adverse effect estimated to occur in up to 40% of patients undergoing chemotherapy, with its incidence increasing in patients being treated with multiple agents. Pharmacists play a pivotal role in the prevention and management of CIPN by recommending evidence-based pharmacologic and non pharmacologic strategies appropriate for the individual patient.Peripheral neuropathy (PN) is a systemic disease characterized by symmetrical, distal damage to the peripheral nerves that negatively impacts patient quality of life (QOL). Prolonged symptoms associated with PN can cause pain, interfere with functional ability (e.g., dressing, driving, house-work), and disrupt emotional health.

ELIGIBILITY:
Inclusion Criteria:

1. Their age will ranging from eight to seventeen years.
2. Children participated in this study will from both sexes.
3. Children receiving chemotherapy as medical treatment protocol
4. All children have polyneuropathy caused by chemotherapy.

Exclusion Criteria:

1. Children with Epilepsy.
2. Children with blood clotting disorder.
3. Children have Open wounds / broken skin
4. Children with severe cardiac disease
5. Uncooperative patients.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction studies (NCS) | nerve conduction velocity for sensory ulnar nerve at day 0
  nerve conduction velocity for sensory ulnar nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory ulnar nerve at day 90
  nerve conduction velocity for sensory ulnar nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sensory median nerve at day 0
  nerve conduction velocity for sensory median nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sensory median nerve at day 90
  nerve conduction velocity for sensory median nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sural nerve at day 0
  nerve conduction velocity for sensory sural nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sural nerve at day 90
  nerve conduction velocity for sensory sural nerve
Nerve conduction studies (NCS) | nerve conduction velocity for motor common peroneal nerve at day 0
  nerve conduction velocity for motor common peroneal nerve
Nerve conduction studies (NCS) | nerve conduction velocity for motor common peroneal nerve at day 90
  nerve conduction velocity for motor common peroneal nerve

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, Ph.D, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Scotte F, Banu E, Medioni J, Levy E, Ebenezer C, Marsan S, Banu A, Tourani JM, Andrieu JM, Oudard S. Matched case-control phase 2 study to evaluate the use of a frozen sock to prevent docetaxel-induced onycholysis and cutaneous toxicity of the foot. Cancer. 2008 Apr 1;112(7):1625-31. doi: 10.1002/cncr.23333. PMID 18286527
- [Background] Hanai A, Ishiguro H, Sozu T, Tsuda M, Yano I, Nakagawa T, Imai S, Hamabe Y, Toi M, Arai H, Tsuboyama T. Effects of Cryotherapy on Objective and Subjective Symptoms of Paclitaxel-Induced Neuropathy: Prospective Self-Controlled Trial. J Natl Cancer Inst. 2018 Feb 1;110(2):141-148. doi: 10.1093/jnci/djx178. PMID 29924336
- [Background] Tsuyuki S, Senda N, Kanng Y, Yamaguchi A, Yoshibayashi H, Kikawa Y, Katakami N, Kato H, Hashimoto T, Okuno T, Yamauchi A, Inamoto T. Evaluation of the effect of compression therapy using surgical gloves on nanoparticle albumin-bound paclitaxel-induced peripheral neuropathy: a phase II multicenter study by the Kamigata Breast Cancer Study Group. Breast Cancer Res Treat. 2016 Nov;160(1):61-67. doi: 10.1007/s10549-016-3977-7. Epub 2016 Sep 12. PMID 27620884
- [Background] Kadakia KC, Rozell SA, Butala AA, Loprinzi CL. Supportive cryotherapy: a review from head to toe. J Pain Symptom Manage. 2014 Jun;47(6):1100-15. doi: 10.1016/j.jpainsymman.2013.07.014. Epub 2013 Nov 7. PMID 24210702

DOCUMENTS (1):
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT04536207/Prot_000.pdf